CLINICAL TRIAL: NCT03030404
Title: Hereditary Gastric Cancer Syndromes: An Integrated Genomic and Clinicopathologic Study of the Predisposition to Gastric Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170043; 17-C-0043
Record Dates: First submitted 2017-01-24; First posted 2017-01-25 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-24

CONDITIONS: Stomach Neoplasms; Stomach Cancer; Gastric Adenocarcinoma and Proximal Polyposis of the Stomach (GAPPS); Hereditary Diffuse Gastric Cancer (HDGC); Familial Diffuse Gastric Cancer
Keywords: Genetics and Germline Mutations; Familial Background; Inherited Cancer Syndrome; Germline Mutation in the CDH1 Gene; Lobular Breast Cancer; Natural History
MeSH Terms: conditions — Stomach Neoplasms; Polyposis, Gastric; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects with suspicious personal or family medical history of gastric cancer or gastric cancer syndrome.

SUMMARY:
Background:

Gastric cancers are cancers of the stomach. Hereditary ones are passed from parent to child. Researchers want to gather data about hereditary gastric cancers. They want to learn about changes these cause in the body and about the genes involved.

Objective:

-To gather data about hereditary gastric cancer.

Eligibility:

* People at least 2 years old with personal or family history with a hereditary gastric cancer.
* People at least 2 years old with gene changes that lead to such cancer or a lesion that may be hereditary.

Design:

* Participants will be screened in a separate protocol.
* Participants will have:

  * Physical exam
  * Medical history
  * Blood tests
  * Scans
  * Photos of skin lesions and other findings
  * Gynecology consultation for women
  * Cheek swab (some participants)
* For some participants, their relatives will be asked to join the study.
* Some participants will be asked to allow the study to get stored tissue samples for relatives who have died.
* Some samples will be sent to outside labs. All personal data will be protected. Samples will be destroyed when the study ends.
* Participants will get the results of genetic testing.
* Participants who cannot come to the NIH clinic may just give a cheek swab and have genetic testing done.
* Some participants will be contacted for more testing.

DETAILED DESCRIPTION:
Background:

An estimated 1-3% of gastric cancer cases occur within a familial background as part of an inherited cancer syndrome.

Hereditary Diffuse Gastric Cancer (HDGC) is the most frequent form of familial gastric cancer and has been linked to a germline mutation in the CDH1 gene.

Gastric Adenocarcinoma and Proximal Polyposis of the Stomach (GAPPS) is a more recently described autosomal dominant syndrome characterized by fundic gland polyposis with antral sparing.

Other germline mutations that predispose to gastric cancer such as SDH (succinate dehydrogenase protein subunits) gene and CTNNA1 (alpha catenin).

Objectives:

Characterize the natural and clinical histories of hereditary gastric cancer syndromes.

Eligibility:

Individuals, and family members, who fulfill clinical criteria for a hereditary gastric cancer syndrome irrespective of previous genetic testing or treatment.

Design:

These rare families will be recruited to genetically confirm diagnosis and study the natural history of hereditary gastric cancers.

Genetic testing will be offered to gain appreciation of the effect of mutations on the relative activity of various germline and somatic mutations.

We will determine if there is a relationship between mutation and disease phenotype.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. An individual, or their family members, with any of the following:

   * Fulfills clinical criteria for Hereditary Diffuse Gastric Cancer (HGDC) syndrome or Gastric Adenocarcinoma and Proximal Polyposis of the Stomach (GAPPS) syndrome.
   * Clinically suspicious personal or family medical history of gastric cancer or gastric cancer syndrome that warrants genetics evaluation.
   * Current diagnosis of gastric cancer and a germline mutation associated with a known cancer syndrome or an associated family history of gastric cancer.
   * Harbors a pathogenic germline mutation known to predispose to gastric cancer.
   * First-degree relatives, regardless of family history or personal history of cancer, with a documented deleterious germline mutation (including but not limited to CDH1, CTNNA1, SDH) known to predispose to gastric tumors.
   * Diagnosis or suspicion of a premalignant or malignant stomach lesion of suspected hereditary etiology.
2. Age >= 2 years and older. Note: Patients under 18 years of age may only participate in research sample collection if the tissue acquisition is performed during a clinically indicated surgical procedure, and the sampling of tissue, blood, saliva or urine collection does not add risk to the clinically indicated procedures.
3. Ability of subject or legally authorized representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals, and family members, who fulfill clinical criteria for a hereditary gastric cancer syndrome irrespective of previous genetic testing or treatment
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Characterization of the natural and clinical histories of hereditary gastric cancer syndromes | 10 years
  Characterization of the natural and clinical histories of hereditary gastric cancer syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Hansford S, Kaurah P, Li-Chang H, Woo M, Senz J, Pinheiro H, Schrader KA, Schaeffer DF, Shumansky K, Zogopoulos G, Santos TA, Claro I, Carvalho J, Nielsen C, Padilla S, Lum A, Talhouk A, Baker-Lange K, Richardson S, Lewis I, Lindor NM, Pennell E, MacMillan A, Fernandez B, Keller G, Lynch H, Shah SP, Guilford P, Gallinger S, Corso G, Roviello F, Caldas C, Oliveira C, Pharoah PD, Huntsman DG. Hereditary Diffuse Gastric Cancer Syndrome: CDH1 Mutations and Beyond. JAMA Oncol. 2015 Apr;1(1):23-32. doi: 10.1001/jamaoncol.2014.168. PMID 26182300
- [Background] Fitzgerald RC, Hardwick R, Huntsman D, Carneiro F, Guilford P, Blair V, Chung DC, Norton J, Ragunath K, Van Krieken JH, Dwerryhouse S, Caldas C; International Gastric Cancer Linkage Consortium. Hereditary diffuse gastric cancer: updated consensus guidelines for clinical management and directions for future research. J Med Genet. 2010 Jul;47(7):436-44. doi: 10.1136/jmg.2009.074237. PMID 20591882
- [Background] van der Post RS, Vogelaar IP, Carneiro F, Guilford P, Huntsman D, Hoogerbrugge N, Caldas C, Schreiber KE, Hardwick RH, Ausems MG, Bardram L, Benusiglio PR, Bisseling TM, Blair V, Bleiker E, Boussioutas A, Cats A, Coit D, DeGregorio L, Figueiredo J, Ford JM, Heijkoop E, Hermens R, Humar B, Kaurah P, Keller G, Lai J, Ligtenberg MJ, O'Donovan M, Oliveira C, Pinheiro H, Ragunath K, Rasenberg E, Richardson S, Roviello F, Schackert H, Seruca R, Taylor A, Ter Huurne A, Tischkowitz M, Joe ST, van Dijck B, van Grieken NC, van Hillegersberg R, van Sandick JW, Vehof R, van Krieken JH, Fitzgerald RC. Hereditary diffuse gastric cancer: updated clinical guidelines with an emphasis on germline CDH1 mutation carriers. J Med Genet. 2015 Jun;52(6):361-74. doi: 10.1136/jmedgenet-2015-103094. Epub 2015 May 15. PMID 25979631
- [Derived] Gallanis AF, Bowden C, Lopez R, Turner J, Fasaye GA, Perati SR, Hernandez JM, Blakely A, Davis JL. Reproductive decision-making and pregnancy in germline CDH1 variant carriers. J Med Genet. 2025 Sep 19;62(10):609-616. doi: 10.1136/jmg-2025-110857. PMID 40541392
- [Derived] Gallanis AF, Gamble LA, Samaranayake SG, Lopez R, Rhodes A, Rajasimhan S, Fasaye GA, Juma O, Connolly M, Joyce S, Berger A, Heller T, Blakely AM, Hernandez JM, Davis JL. Costs of Cancer Prevention: Physical and Psychosocial Sequelae of Risk-Reducing Total Gastrectomy. J Clin Oncol. 2024 Feb 1;42(4):421-430. doi: 10.1200/JCO.23.01238. Epub 2023 Oct 30. PMID 37903316
- [Derived] Green BL, Gamble LA, Diggs LP, Nousome D, Patterson JC, Joughin BA, Gasmi B, Lux SC, Samaranayake SG, Miettinen M, Quezado M, Hernandez JM, Yaffe MB, Davis JL. Early Immune Changes Support Signet Ring Cell Dormancy in CDH1-Driven Hereditary Diffuse Gastric Carcinogenesis. Mol Cancer Res. 2023 Dec 1;21(12):1356-1365. doi: 10.1158/1541-7786.MCR-23-0122. PMID 37707375
- [Derived] Gamble LA, Lopez R, Rajasimhan S, Samaranayake SG, Bowden C, Famiglietti AL, Blakely AM, Jha S, Ahlman MA, Davis JL. Micronutrient Supplementation and Bone Health After Prophylactic Total Gastrectomy in Patients With CDH1 Variants. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2635-2642. doi: 10.1210/clinem/dgad137. PMID 36950857
- [Derived] Passi M, Gamble LA, Samaranayake SG, Schueler SA, Curtin BF, Fasaye GA, Bowden C, Gurram S, Quezado M, Miettinen M, Koh C, Heller T, Davis JL. Association of CDH1 Germline Variants and Colon Polyp Phenotypes in Patients with Hereditary Diffuse Gastric Cancer. Gastro Hep Adv. 2023;2(2):244-251. doi: 10.1016/j.gastha.2022.10.006. Epub 2022 Oct 28. PMID 36776716
- [Derived] Gamble LA, Grant RRC, Samaranayake SG, Fasaye GA, Koh C, Korman L, Asif B, Heller T, Hernandez JM, Blakely AM, Davis JL. Decision-making and regret in patients with germline CDH1 variants undergoing prophylactic total gastrectomy. J Med Genet. 2023 Mar;60(3):241-246. doi: 10.1136/jmg-2022-108733. Epub 2022 Jul 11. PMID 35817563
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0043.html